CLINICAL TRIAL: NCT00799513
Title: A Phase II Trial to Evaluate the Safety and Activity of Single-agent Lenalidomide Given as Maintenance Therapy After Response to Second-line Therapy in Patients With Relapsed DLBCL, Not Eligible for High-dose Chemotherapy and ASCT (Autologous Stem-Cell Transplantation)
Brief Title: Trial on Lenalidomide Given as Maintenance Therapy for Relapsed Diffuse Large B Cell Lymphoma
Acronym: RV-NHL-PI351
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Andrés José Maria Ferreri, Unit Head, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-003729-18; 2008-003729-18 (EudraCT Number)
Record Dates: First submitted 2008-11-20; First posted 2008-12-01 (Estimated); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Lenalidomide; revlimid; large B-cell lymphoma; relapse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): single-agent lenalidomide 25 mg once daily for 21 days out of 28, as maintenance treatment after the end of second-line chemotherapy until progression of disease.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — single-agent lenalidomide 25 mg once daily for 21 days out of 28, as maintenance treatment after the end of second-line chemotherapy until progression of disease.
  Other Names: Revlimid

SUMMARY:
This phase II multi-institutional trial will explore the safety and efficacy of lenalidomide monotherapy given as maintenance therapy following salvage chemo-immunotherapy in patients with relapsed or refractory chemosensitive diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
Patients older than 65 years or younger but not eligible to high-dose chemotherapy and autologous stem cell transplantation with biopsy-proven diffuse large B-cell lymphoma relapsed to previous combination chemotherapy regimen ± rituximab, who achieved at least a partial response to second-line chemotherapy (ICE or DHAP/DHAOx ((D)examethasone (H)igh-dose (A)ra-C - cytarabine (P)latinol (cisplatin)) or MINE (Mesna Ifosfamide Mitoxantrone Etoposide) regimen) + rituximab will receive single-agent lenalidomide 25 mg once daily for 21 days out of 28, as maintenance treatment until progression of disease. Dose reductions of study drug will be made in case of adverse events when reported as correlated and when clinically appropriate.

One-year progression free survival (PFS) will be the primary endpoint and overall survival, response rate and toxicity will be the secondary endpoints. With the null hypothesis (P0) of 1-year PFS of 30%, this study will consider a satisfactory efficacy of lenalidomide worth of further investigation a P1 corresponding to a 1-yr PFS of 50% (that is an absolute increase of 20% in terms of 1-yr progression-free survival). Considering a standard type I error (α) of 0,05 and a power of 80% (Type 2 error of 20%) 47 patients will be necessary for the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Age < 65 but not eligible to high-dose chemotherapy and autologous stem cell transplantation
* Biopsy-proven DLBCL relapsed to previous combination chemotherapy regimen ± rituximab
* PR (Partial Response) or CR (Complete Response) to second-line chemotherapy (ICE or DHAP/DHAOx or MINE regimen) + rituximab
* ECOG (Eastern Cooperative Oncology Group) performance status score < 4
* Female of childbearing potential (FCBP) must demonstrate to practice a proper contraception to avoid any pregnancy risk during the study and at least 28 days after the discontinuation of the study
* Male subjects must agree to practice a proper contraception during any sexual contact with females childbearing potential

Exclusion Criteria:

* CNS (Central Nervous System) involvement
* Prior ASCT
* TTP (Time To Progression) <6 months after first-line therapy
* Use of experimental drugs during second-line salvage chemotherapy
* Severe concomitant illnesses / medical conditions (e.g. impaired respiratory and/or cardiac function, uncontrolled diabetes mellitus )
* Active infectious disease
* HIV, HBV (Hepatitis B Virus) or HCV (Hepatitis C Virus) - positivity
* Impaired liver function (Bilirubin >2 x upper normal limit; ALT (alanine aminotransferase) /AST (aspartate aminotransferase) /GGT (γ-glutamyltransferase) > 3 x upper normal limit) at one month from salvage chemotherapy conclusion
* Impaired renal function (creatinine clearance <50 ml/min) at one month from salvage chemotherapy conclusion
* Absolute neutrophil count (ANC) <1000/microL
* Platelet count <75.000 /mm3
* Hemoglobin <9 g/dL
* Non-co-operative behaviour or non-compliance
* Psychiatric diseases or conditions that might impair the ability to give informed consent
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrés J. Ferreri, MD, Study Chair — San Raffaele Scientific Institute
Locations (1):
- San Raffaele Scientific Institute, Milan, Italy

REFERENCES:
- [Derived] Ferreri AJ, Sassone M, Zaja F, Re A, Spina M, Rocco AD, Fabbri A, Stelitano C, Frezzato M, Rusconi C, Zambello R, Couto S, Ren Y, Arcari A, Bertoldero G, Nonis A, Scarfo L, Calimeri T, Cecchetti C, Chiozzotto M, Govi S, Ponzoni M. Lenalidomide maintenance in patients with relapsed diffuse large B-cell lymphoma who are not eligible for autologous stem cell transplantation: an open label, single-arm, multicentre phase 2 trial. Lancet Haematol. 2017 Mar;4(3):e137-e146. doi: 10.1016/S2352-3026(17)30016-9. Epub 2017 Feb 17. PMID 28219694
- [Derived] Vose JM, Habermann TM, Czuczman MS, Zinzani PL, Reeder CB, Tuscano JM, Lossos IS, Li J, Pietronigro D, Witzig TE. Single-agent lenalidomide is active in patients with relapsed or refractory aggressive non-Hodgkin lymphoma who received prior stem cell transplantation. Br J Haematol. 2013 Sep;162(5):639-47. doi: 10.1111/bjh.12449. Epub 2013 Jul 9. PMID 23834234

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide
Started | 48
Completed | 46
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 39
Age, Continuous [Median (Full Range); unit: years] | 72 [34 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 46
Relapse Status [Count of Participants; unit: Participants]
  First | 33
  Second | 13
Previous Lines for Diffuse Large B Cell Lymphoma (DLBCL) treatment [Count of Participants; unit: Participants] — The different treatments for the medical condition used before the trial
  Participants
    Rituximab Cyclophosphamide Hydroxydaunorubicin Oncovin Prednisone.(R-CHOP) | 38
    Rituximab+methotrexate+Adriamycin+cyclophosphamide+Oncovin+prednisone+bleomycin(R-VACOP-MACOP-B | 8
Previous ASCT (Autologous Stem-Cell Transplantation) [Count of Participants; unit: Participants] | 6
Eastern Cooperative Oncology Group (ECOG) Performance Score >=1 [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group is a 0 to 5 scale which define health status 0 is perfectly healthy 5 is death
  Participants | 18
International Prognostic Index [Count of Participants; unit: Participants] — The International Prognostic Index (IPI) is a clinical tool developed by oncologists to aid in predicting the prognosis of patients with aggressive non-Hodgkin's lymphoma:
  Low risk (0-1 points) - 5-year survival of 73% Low-intermediate risk (2 points) - 5-year survival of 51% High-intermediate risk (3 points) - 5-year survival of 43% High risk (4-5 points) - 5-year survival of 26%
  Participants
    Low- 5-year survival of 73% | 8
    Low-Intermediate- 5-year survival of 51% | 21
    High-Intermediate- 5-year survival of 43% | 12
    High- 5-year survival of 26% | 5
Advanced stage of disease [Count of Participants; unit: Participants] | 35
Increased LDH (lactate dehydrogenase) serum level [Count of Participants; unit: Participants] | 21
Systemic symptoms (B status) [Count of Participants; unit: Participants] | 5
Extranodal disease [Count of Participants; unit: Participants] | 29
Bone marrow infiltration [Count of Participants; unit: Participants] | 6
Hepatitis viral infection [Count of Participants; unit: Participants]
  Hepatitis B Virus | 7
  Hepatitis C Virus | 2
  Both | 3
  None | 34
Salvage chemoimmunotherapy [Count of Participants; unit: Participants]
  High-dose Cytarabine-based: DHAP | 10
  High-dose Cytarabine-based:DHAOx | 10
  High-dose Cytarabine-based: ESHAP | 3
  High-dose Ifosfamide-based: ICE | 8
  Anthracycline-based: CHOP | 6
  Bendamustine | 5
  Gemcitabine-oxaliplatin | 4
Response at time of trial registration [Count of Participants; unit: Participants]
  Complete remission | 26
  Partial remission | 20

OUTCOME MEASURES:

1. Primary Outcome: 1-year Progression-free Survival
Description: It is defined as the number of participants alive after 1 year from enrolment to progression or relapse of lymphoma (if post-induction disease status was PR (Partial Response) or CR (Complete Response), respectively). Patients alive at last follow-up will be censored.
Time Frame: 1-year
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 46
Participants | 31

2. Secondary Outcome: Progression Free Survival
Description: Secondary measures to describe long term outcome of treatment
  -Progression free survival It is defined as the number of participants, on a 5 yrs follow up, free from disease progression
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 46
Participants | 25

3. Secondary Outcome: Progression
Description: Progression It is defined as the number of participants with disease recurrence observed on a 5 yrs follow up.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 46
Participants | 21

4. Secondary Outcome: Duration of Response
Description: Secondary measures to describe long term outcome of treatment
  * Duration of response It is defined as the number of participants experiencing a PFS (Progression Free Survival) from study therapy longer than previous line of treatment
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 46
Participants | 29

5. Secondary Outcome: Overall Survival
Description: Secondary measures to describe long term outcome of treatment
  -Overall survival It is defined as the number of participants alive at 5ys from enrolment (death for any cause). Patients alive at last follow-up will be censored.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 46
Participants | 26

ADVERSE EVENTS:
Time Frame: 5 years
Description: Definition per International Conference on Harmonization (ICH)
Arm/Group | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 22/48
Serious Adverse Events (participants affected / at risk) | 12/48
Other Adverse Events (participants affected / at risk) | 7/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=48)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
diarrhea (Gastrointestinal disorders) | 2 (2)
melena (Gastrointestinal disorders) | 1 (1)
stroke (Vascular disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
Herpes voster virus (Infections and infestations) | 1 (1)
intestinal infraction (Gastrointestinal disorders) | 1 (1)
meningitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=48)
Neutropenia G3+ (Blood and lymphatic system disorders) | 7 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT00799513/Prot_SAP_000.pdf